CLINICAL TRIAL: NCT02628288
Title: COmplex Bifurcation Lesions: a RAndomized Comparison Between the AXXESS Device in Combination With Absorb BVS, and Modified T Stenting With Absorb BVS: an OCT Study.
Brief Title: COmplex Bifurcation PCI: AXXESS Device + Absorb BVS, vs Modified T Stenting With Absorb BVS
Acronym: COBRAII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-57892
Record Dates: First submitted 2015-11-17; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCI with Axxess device + AbsorB BVS (Active Comparator): Bifurcation lesion will be treated percutaneously by performing coronary stenting with AXXESS device and additional Absorb BVS.
  Interventions: Device: Coronary Bifurcation PCI
- PCI with Modified T with Absorb BVS (Active Comparator): Bifurcation lesion will be treated percutaneously by performing coronary stenting with a modified T stenting technique using Absorb BVS.
  Interventions: Device: Coronary Bifurcation PCI

INTERVENTIONS:
Device: Coronary Bifurcation PCI — In one group, the coronary bifurcation lesion will be treated (Coronary bifurcation PCI) with the Axxess device + Absorb BVS. In the other group, the coronary bifurcation lesions will be treated(Coronary bifurcation PCI) by modified T stenting using Absorb BVS.

SUMMARY:
Comparison of healing responses after treatment of complex bifurcation lesions with a dedicated bifurcation device (Axxess™ Biolimus Eluting Coronary Bifurcation Stent System + Absorb BVS in the distal branches) versus the Modified T stenting technique using Absorb BVS: an optical coherence tomography (OCT) analysis.

DETAILED DESCRIPTION:
This is a prospective single center randomized clinical trial with baseline OCT and clinical, angiographic and OCT follow-up at thirty months. Patients with true and complex coronary bifurcation lesions are randomly assigned to treatment with the dedicated Axxess biolimus-eluting bifurcation stent in the proximal main vessel (MV) and additional Absorb everolimus-eluting BVS in the branches versus a modified T technique using Absorb BVS only. The primary endpoint is changes in minimal luminal area assessed with OCT from baseline to 30 months in pre-specified bifurcation segments. The main aims are to assess acute performance and to compare long-term vessel healing with optical coherence tomography, and clinical and angiographic outcome after treatment of complex bifurcation lesions with a dedicated stent with additional Absorb Bioabsorbable scaffolds (BVS) versus a modified T stenting technique with Absorb BVS.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years
2. The subject has stable or unstable angina pectoris, or a positive functional study for ischemia.
3. The subject is eligible for PCI, and is an acceptable candidate for coronary artery bypass surgery.
4. The subject is male, or if female, has no childbearing potential or has had a negative urine or serum pregnancy test within 7 days of the index procedure and has no intention to become pregnant within a year of the procedure.
5. The subject has signed the informed consent prior to the procedure, and agrees to comply with the follow up requirements.
6. Patients with a de novo and true coronary bifurcation lesion (Medina classification (1,1,1), (1,0,1) or (0,1,1)) or any other anatomical presentation requiring a double stent technique by judgment of the operator.
7. Coronary artery with proximal parent vessel reference diameter of 2.75 - 3.75 mm and a branch vessel diameter of ≥ 2.25 mm (by visual estimate).
8. The lesion must be at least 50% diameter stenosis within either the MB or SB (by visual estimate).
9. Regarding lesion length: lesion should be able to be covered by 2 Absorb BVS in a Modified T-stenting technique, or by a combination of maximally 1 AXXESS and 2 Absorb BVS (by visual estimate).
10. The side branch ostium is located at least 10 mm from the left main coronary artery (by visual estimate).
11. The angle between the sidebranch and the parent vessel is less than 70°(by visual estimate).

Exclusion Criteria:

1. Left ventricular ejection fraction of < 30%
2. Impaired renal function (serum creatinine > 2.0 mg/dl)
3. Previous and/or planned brachytherapy of target vessel
4. Known allergies to antiplatelet, anticoagulation therapy, contrast media, biolimus or everolimus, nickel, titanium or poly-D,L-lactic Acid.
5. Pregnant and/or breast-feeding females or females who intend to become pregnant (pregnancy test required)
6. Patients with a life expectancy of less than three years
7. Patient currently enrolled in other investigational device or drug trial of which the primary endpoint timing has not been reached and potentially interferes with the outcome of either of both trials
8. Patient not able or willing to adhere to follow-up visits
9. Patients who intend to have a major surgical intervention within 12 months of enrolment in the study.
10. Patients who previously participated in this study.
11. Subject has experienced an acute myocardial infarction 72 hours prior to the index procedure, as defined either by the presence of a new Q-wave in 2 or more contiguous leads, or by a CK greater than two times site upper reference limit (URL) with presence of creatine Kinase-MB ( CKMB) greater than the site URL.
12. Creatinine Kinase (CK) greater than two times URL with presence of CKMB greater than the site URL at the time of procedure.
13. The subject has suffered a stroke or transient ischemic neurological attack or cerebrovascular accident within the past six months, or has any known intracranial mass, arteriovenous malformation, aneurysm or other intracranial pathology
14. The subject has experienced a significant gastrointestinal or genitourinary bleed within the past six months, or has had any active bleeding within two months.
15. The subject is taking warfarin or NOAC, will need to take warfarin or novel oral anticoagulants (NOAC) post procedure, or has an international normalised ratio (INR) > 1.4.
16. Planned revascularization within 1 year after index procedure.
17. The target vessel contains intraluminal thrombus.
18. The target lesion is located in the left main coronary artery
19. Lesion of the left main trunk > 50%, unprotected
20. The subject has another lesion within the target vessel parent or side branch requiring treatment besides the bifurcation lesion
21. The subject has had prior PCI to the target lesion, including a 5mm zone proximal and distal to the lesion
22. The target lesion shows angiographic evidence of severe calcification or tortuosity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-03 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Changes in minimal luminal area in 4 pre-specified bifurcation segments (Proximal mainbranch (MB) segment; Bifurcation segment; Ostial distal MB segment; Ostial side-branch (SB segment), assessed with OCT, from baseline to 30 months. | 30 months

SECONDARY OUTCOMES:
Acute strut apposition following index PCI (baseline OCT) | 30 months
Cumulative major adverse cardiac events (MACE) rate (cardiac death, myocardial infarction, clinically driven TLR) at 1, 6 and 12 months and annually for 5 years from the procedure date. | 1 month, 6 months, 1,2,3,4,5 years
Quantitative coronary angiography (QCA) Minimal Lumen Diameter before and after PCI, and at 30 months | 24 hours and at 30 months
Device success, defined as deployment of the assigned stents without system failure or device-related complication | 24 hours
Presence of thrombus on final OCT pullback following index PCI | 24 hours
- Assessment of the integrity of the Absorb BVS following completion of index PCI using 3D OCT. | 24 hours
Minimal lumen area at baseline and follow-up in the other 6 pre-specified bifurcation segments (Proximal edge segment; Proximal MB segment; Distal MB segment; Distal MB edge segment; SB segment: Distal SB edge segment) | 24 hours and 30 months
Changes in minimal luminal area in all 10 pre-specified bifurcation segments, assessed with OCT, from baseline to 30 months. | 24 hours and 30 months
Percent struts malapposed in the Axxess stent at 30 months post procedure | 30 months
Percent struts uncovered in the Axxess stent at 30 months post procedure | 30 months
Target vessel failure (TVF), defined as the combination of cardiac death, target vessel myocardial infarction, or clinically driven target lesion revascularisation (TLR) | 1 month, 6 months, 1,2,3,4,5 years
Stent thrombosis at 24h, 1 month, 12 months and yearly thereafter (up to 5y) | 1 month, 6 months, 1,2,3,4,5 years
Target lesion revascularisation (TLR) at 1, 6, 12 months and yearly thereafter (up to 5y) | 1 month, 6 months, 1,2,3,4,5 years
Target vessel revascularisation (TVR) at at 1, 6, 12 months and yearly thereafter (up to 5y) | 1 month, 6 months, 1,2,3,4,5 years
All-cause death, cardiac death, non-TVR, any revascularization at 1, 6, 12 months and yearly thereafter (up to 5y) | 1 month, 6 months, 1,2,3,4,5 years
Acute gain following index PCI | 24 hours
Late Lumen Loss (in-stent) at 30 months | 30 months
Binary in-stent/scaffold restenosis at 30 months | 30 months
Binary in-segment restenosis at 30 months | 30 months
Binary in-bifurcation restenosis (stent and segment) at 30 months | 30 months
Lesion success, defined as attainment of <50% residual stenosis of the target lesion using any percutaneous method | 24 hours
Procedure success, defined as lesion success without the occurrence of MACE during the hospital stay. | 24 hours
Analysis of the vasoreactivity (Vasomotor testing, using vasodilatory response to acetylcholine (Ach) in all patients) of the bifurcation segments previously stented/scaffolded. | 30 months
Procedure duration from randomization to final angiogram (before final OCT) | 24 hours
Contrast usage from randomization to final angiogram (before final OCT) | 24 hours
Radiation from randomization to final angiogram (before final OCT) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bennett, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Department of Cardiovascular Disease, University Hospitals Leuven, Leuven, Belgium